CLINICAL TRIAL: NCT04591262
Title: A PHASE 1, OPEN LABEL, 2-PERIOD, FIXED SEQUENCE, STUDY TO ASSESS THE MASS BALANCE, ABSOLUTE BIOAVAILABILITY OF 14C PF 06826647 IN HEALTHY MALE PARTICIPANTS
Brief Title: A Study To Asses Mass Balance And Absolute Bioavailability Of 14C PF-06826647 In Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C2501006
Record Dates: First submitted 2020-09-09; First posted 2020-10-19 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: ADME, Mass Balance, Absolute Bioavailability, AMS
MeSH Terms: interventions — ropsacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PF-06826647 600 mg PO>PF-06826647 600 mg PO+100 ug IV (Experimental): PF-06826647 600 mg single dose in Period 1 followed by PF-06826647 600 mg PO and IV infusion of 100 ug of PF-06826647 in Period 2.
  Interventions: Drug: 14C-PF-06826647-LR 600 mg PO; Drug: PF-06826647 600 mg PO; Drug: 14C-PF-06826647 100 ug IV

INTERVENTIONS:
Drug: 14C-PF-06826647-LR 600 mg PO — 14C-PF-06826647-LR 600 mg with 300 nCi orally as extemp prep
Drug: PF-06826647 600 mg PO — Unlabeled PF-06826647 600 mg
Drug: 14C-PF-06826647 100 ug IV — 14C-PF-06826647 100 ug IV

SUMMARY:
The purpose of the study is to determine the metabolism and excretion following a single oral administration of 14C-PF-06826647-LR (14C labelled PF-06826647 with lower radioactivity per mass unit) in fed conditions. This information will enable assessment of clearance mechanisms of PF-06826647 as well as identify metabolites. In addition, this study will determine absolute bioavailability of PF-06826647 and understand intravenous (IV) pharmacokinetic (PK).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male participants must be 18 to 55 years of age, inclusive.
* Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, including BP and pulse rate measurement, laboratory tests, and 12 lead ECG.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI of 17.5 to 30 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of irregular bowel movements including irritable bowel syndrome or frequent episodes of diarrhea or constipation defined by less than 1 bowel movement on average per 2 days or lactose intolerance.
* Participants who currently use or have formerly used (within 6 months of dosing) tobacco or nicotine containing products.
* Total 14C radioactivity measured in plasma exceeding 11 mBq/mL.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in urine and feces together expressed as percent of total oral radioactive dose | Up to Day 14

SECONDARY OUTCOMES:
Number of Participants With Laboratory Test Values of Potential Clinical Importance | Up to Day 28
  Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance.
Number of participants with abnormal ECG | Up to Day 28
  Criteria for ECG abnormalities: maximum PR interval >=300 milliseconds (msec) and maximum increase PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 msec and Pctchg>=50% for baseline value of <=200 msec for PR interval, maximum QRS interval >=140 msec and a maximum IFB: Pctchg>=50%, maximum QTCF interval (Fridericia's Correction) of 450 msec to <480 msec, 480 msec to <500 msec or >=500 msec and a maximum change of <=30change<60 or >=60 msec from baseline.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Up to Day 28
  Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, respiratory rate, radial pulse and body temperature.
The ratio of dose normalized AUCinf of PF-06826647 and 14C-PF-06826647 | 0 hours to 96 hours
  The ratio of dose normalized AUCinf of PF-06826647 (LCMS) and 14C-PF-06826647 (AMS). AUCinf= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time . It is obtained from AUC (0 - t) plus AUC (t - ∞).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - PRA Health Sciences, Groningen
  - PRA Health Sciences Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2501006